CLINICAL TRIAL: NCT03524625
Title: Sensitivity and Specificity of a Mobile Lead-one ECG Like Device for the Detection of Atrial Fibrillation (AF)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 1806643
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrial Fibrillation(AF) is one of the most common abnormal heart rhythms and approximately 3% of the general population have AF. The prevalence increases with age of the population and is increased in people with diabetes, hypertension and those who are overweight. AF is a major risk factor for stroke; people with AF are five times more likely to suffer an ischaemic stroke; however this can be reduced significantly with appropriate interventions which depends on detection of the abnormal rhythm. Although the National Institute of Health and Care Excellence (NICE) currently recommends screening patients with symptoms of AF, including syncope, heart palpitations, and chest discomfort, as well as patients who have suffered a stroke or heart attack, many patients remain symptomless and are not managed for their increased stroke risk. Guidelines for AF screening include manual palpation of a peripheral pulse, followed up by an ECG for patients who have an irregular pulse. Although almost all patients with AF have an irregular pulse, only about 12 in 100 patients with an irregular pulse have AF. Use of an improved screening tool for AF could both cut down the number of people undergoing unnecessary ECGs, and also lead the way for a wider screening programme for AF. The aim of this study is to investigate the sensitivity and specificity of a new ECG like device for the detection of AF, the Plessey imPulse. Participants referred or admitted to secondary care with stroke symptoms and other indicators of increased prevalence of AF will be recruited. Participants will undergo three methods of AF screening, a peripheral pulse, a lead-one like ECG using the imPulse device, and the gold-standard for AF detection, a 12-lead ECG. By comparing to the ECG results specificity and sensitivity will be established for both methods in this population.

ELIGIBILITY:
Inclusion Criteria:

Patients with AF or suspected AF referred or admitted to hospital (secondary care setting). Able to hold the impulse device with both hands. Able to give informed consent.

Exclusion Criteria:

Patients who are unable to give informed consent either through lack of capacity or lack of ability to understand study documentation. Patients who are unable to hold the impulse device for 2mins. Presence of artificial pacemaker or cardioverter defibrillator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to secondary care to investigate stroke symptoms at the Stroke Clinic will be the primary target for recruitment. However, to enrich the sample with more confirmed AF patients, admitted secondary care patients will also be recruited. Once the sensitivity and specificity has been established in this AF enriched cohort a larger study (in the primary care setting) is planned.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the Plessey imPulse lead-I ECG like device for detecting AF. | 6months
  The primary aim of this study is to evaluate the diagnostic accuracy of the Plessey imPulse lead-I ECG like device for detecting AF.
  Objectives:
  * Assess sensitivity
  * Assess specificity
  * Assess positive predictive value
  * Assess negative predictive value In addition to providing estimates of diagnostic performance of the impulse device, the results of this study are intended to inform the trajectory to undertake a follow up study to confirm diagnostic performance in primary care practice setting and its acceptability and clinical utility.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Clark, MD, Principal Investigator — University Of Exeter Medical School
Locations (1):
- Royal Devon and Exeter NHS Trust, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Research data in digital format in a clinical trial data base and on secure University of Exeter servers will be kept for 5 years to allow time to analyse the results and publish the research.